CLINICAL TRIAL: NCT02479672
Title: Comparison of the VividTrac® Videolaryngoscope to Direct Laryngoscopy in Adults Under Manual Inline Stabilization
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was never started.
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Mathew Malkin, MD, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 5150229
Record Dates: First submitted 2015-06-17; First posted 2015-06-24 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Endotracheal Intubation
Keywords: breathing tube placement; VideoTrac® laryngoscope; direct laryngoscopy
MeSH Terms: interventions — Laryngoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VividTrac video laryngoscope (Active Comparator): VividTrac® Videolaryngoscope, A device for endotracheal intubation
  Interventions: Procedure: Manual Inline Stabilization; Device: VividTrac®
- Direct laryngoscopy (Active Comparator): Direct laryngoscopy, A device for endotracheal intubation
  Interventions: Device: laryngoscopy; Procedure: Manual Inline Stabilization

INTERVENTIONS:
Device: laryngoscopy — Placement of endotracheal tube. If successful intubation does not occur after the first attempt at laryngoscopy, airway equipment used in further attempts will be selected at the discretion of the attending anesthesiologist.
  Arms: Direct laryngoscopy
Procedure: Manual Inline Stabilization — Manual immobilization of Patient's neck with intention to minimize movement from baseline position
Device: VividTrac®
  Arms: VividTrac video laryngoscope

SUMMARY:
This is a prospective randomized clinical study to be performed in adult patients ages 18 and older who are undergoing surgical procedures requiring endotracheal intubation. Adult patients will be randomized to either the VideoTrac® laryngoscope or direct laryngoscopy and the time to intubation will be compared and recorded. Patients in both treatment arms will receive manual inline stabilization. The study hypothesis is that the time to endotracheal intubation will be decreased in the VividTrac® video laryngoscope group when compared to direct laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be 18 years old and older requiring endotracheal intubation

Exclusion Criteria:

* Patients with increased pulmonary risk;
* Prior documentation of difficult endotracheal intubation;
* elevated intracranial pressure;
* those who lack legal representative consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Time to Intubation | day of surgery
  Time frame being assessed will begin at the time of mouth opening and end with the removal of the tip of laryngoscope blade from the patient's mouth after successful endotracheal intubation.